CLINICAL TRIAL: NCT06607822
Title: Development and Validation of a Large Language Model-based Myopia Assistant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSEARS20240229009
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Myopia; Large Language Model
Keywords: Myopia; Large language model; Assistance
MeSH Terms: conditions — Myopia; Helping Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient-centered assistant system (Experimental): Participants engaged in the outpatient clinic visit procedure with a patient-centered assistant system based on Large-Language Model (LLM) for 10 minutes.
  Interventions: Device: A patient-centered assistant system based on Large-Language Model (LLM)
- Control group (No Intervention): Participants engaged in the outpatient clinic visit procedure without the support of patient-centered assistant system based on Large-Language Model (LLM) or any similar artificial intelligence assistance for 10 minutes.

INTERVENTIONS:
Device: A patient-centered assistant system based on Large-Language Model (LLM) — Participants will engage in a 10-minute medical consultation using LLM model interface embedded in a tablet device before their regular face-to-face consulation with physicians. During the trials, participants could engage in free conversations covering aspects including risk factors, symptoms, diagnosis, examinations, treatment, advice and caution, etc. Participants who have completed the ophthalmic imaging examination will be asked to input results into the assistant model to generate structured reports.
  Arms: Patient-centered assistant system

SUMMARY:
Myopia is a rapidly growing global health concern, and there is an urgent need for advanced tools that can facilitate personalized healthcare strategies. Artificial intelligence (AI)-based solutions, such as large language models, offer robust tools for ophthalmic healthcare. In this study, investigators aim to validate a patient-centered Large Language Model (LLM)-based Myopia Assistant System with the following key objectives: 1) evaluate the ability of the LLM models to generate high-level reports and help self-evaluation of myopia for patients in primary care; 2) evaluate its performance in answering evidence-based medicine-oriented questions and improving overall satisfaction within clinics for myopic patients.

DETAILED DESCRIPTION:
Myopia is a rapidly growing global health concern particularly affecting children and adolescents. The progression of myopia can lead to severe complications such as myopic macular degeneration, significantly impacting visual acuity and quality of life. With the rising prevalence of myopia, there is an urgent need for advanced tools that can facilitate personalized healthcare strategies. Artificial intelligence (AI)-based solutions, such as large language models, offer robust tools for ophthalmic healthcare. Nevertheless, their effectiveness and safety in real clinical environments have not been fully explored.

In this study, investigators aim to validate a patient-centered Large Language Model (LLM)-based Myopia Assistant System with the following key objectives: 1) evaluate the ability of the LLM models to generate high-level reports and help self-evaluation of myopia for patients in primary care; 2) evaluate its performance in answering evidence-based medicine-oriented questions and improving overall satisfaction within clinics for myopic patients. The findings of this study will provide valuable insights for the application of the GPT model in the healthcare field, making a significant contribution to improving the accessibility and quality of medical services.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient participants aged 6 to 75.
2. Participants who undergo ophthalmic examinations for medical purposes.
3. Participants who can produce clear ophthalmic images in both eyes.
4. No prior experience in research involving digital medicine
5. Agree to participate in this study with written informed consent

Exclusion Criteria:

1. Participants who are reluctant to participate in this study
2. Participants who are unable to understand the study.
3. Participants who have recently undergone ocular surgery or those with severe ocular conditions that may affect the interpretation of imaging results related to myopia evaluation (e.g., severe vitreous hemorrhage, cataracts, corneal leukoma, etc.) will be excluded from the study.
4. Participants with poor quality of ophthalmic images, including blurriness, artifacts, underexposure, or overexposure.
5. Other unsuitable reasons determined by the evaluators.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Satisfaction level | Immediately after the outpatient clinic visit procedure
  Participants satisfaction level of the clinical experience with or without the use of a patient-centered assistant system based on a large language model (LLM) was assessed. The total satisfaction score was reported using the questionnaire (Patient User Satisfaction Scale), which evaluated the participant satisfaction with the clinical experience and the effectiveness of resolving their own issues. The questionnaire was measured on a 5-point Likert scale, where 1 represents strongly disagree; and 5 represents strongly agree; with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Whether participants adopt the myopia management advice from the physician | Immediately after the outpatient clinic visit procedure
  It is a binary outcome that assesses whether participants follow the recommendations from the physician for myopia management. It focuses on whether participants implement the prescribed treatments or interventions provided to control or manage their myopia.

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, M.D, Ph.D, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided